CLINICAL TRIAL: NCT02152241
Title: Long-term Functional Outcome of Children With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: H2014:155
Record Dates: First submitted 2014-05-26; First posted 2014-06-02 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; Crohn; Colitis; Function
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with IBD: Adult patients with IBD diagnosed during childhood

SUMMARY:
Inflammatory bowel diseases (IBD) are group of immune system disorders characterized by a chronic course with remission and relapses. Canada is one of the countries with the highest prevalence and incidence rates of IBD with 25% of patients present in children and adolescents.

As with any chronic illness, IBD diagnosed early in life has a significant impact on the physical, emotional and social development of those affected. Consequently, it is logical to speculate that patients with IBD may not do as well in education levels or employment status attained compared to their peers without IBD. If this were the case, then interventions could begin in childhood to better prepare patients with IBD for the challenges of living with a chronic disease. Alternatively, if it is shown that they reach comparable social or employment milestones as adults compared to unaffected peers then this would be enormously reassuring to children and their parents.

Properly designed studies to help in defining more appropriate interventions to these patients are needed.

The proposed study includes circulating a survey to evaluate the functioning level of adult patients with IBD who were diagnosed during their childhood. The participants will be asked a series of questions regarding their highest level of educational achievement, the nature of their current employment, and their current marital status. The question format will parallel that of the Canadian Community Health Survey from which data from an age matched healthy adult Manitobans will be extracted and used as another control group. Responses will be analysed for any possible differences between these groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who were initially diagnosed with IBD in childhood or adolescence (diagnosis was made < age of 18 years) and who were followed by the Section of Pediatric Gastroenterology at the Winnipeg Children's Hospital from 1974 - 2009.

Exclusion Criteria:

* Patients in whom the diagnosis of IBD was not fully established following the current North American Society of Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN) guidelines for diagnosing IBD i.e. had clinical, radiologic and endoscopic evidence of IBD (2).
* Control participants with other chronic debilitating diseases (e.g. malignancy, rheumatoid arthritis, multiple sclerosis, etc..) that may affect quality of life and functional outcome

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participant population will be comprised of adult patients who were initially diagnosed with IBD in childhood or adolescence (diagnosis was made < age of 18 years) and who were followed by the Section of Pediatric Gastroenterology at the Winnipeg Children's Hospital from 1974 - 2009.
  Controls: age and sex-matched control group will be generated using the Canadian Community Health Survey (CCHS) 2012 (16) with access through the local Research and Data Centre (RDC).
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Functional outcome (highest level of education attained and current occupation) of those with IBD compared to age and sex-matched healthy adult Manitobans | 12 months
  The highest level of education attained and current occupation will be obtained from participants using structured questionnaire (non-validated interview questionnaire) e.g.
  Employed: Y N If No, Unemployed Y N, Disabled Y N , Homemaker Y N Student Y N, Retired Y N Is the cause of not working disease-related Y N

SECONDARY OUTCOMES:
Functional outcome of patients with Crohn's disease (CD) versus those with ulcerative colitis (UC) | 12 months
  The same structured questionnaire tool will be used. Data will be collected on the highest level of education achieved and the current occupation including any periods of unemployment and if this is disease-related or not

CONTACTS AND LOCATIONS:
Overall Officials: Wael El-Matary, MD, Principal Investigator — Associate Professor, Univeristy of Manitoba
Locations (1):
- HSC, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] El-Matary W, Dufault B, Moroz SP, Schellenberg J, Bernstein CN. Education, Employment, Income, and Marital Status Among Adults Diagnosed With Inflammatory Bowel Diseases During Childhood or Adolescence. Clin Gastroenterol Hepatol. 2017 Apr;15(4):518-524. doi: 10.1016/j.cgh.2016.09.146. Epub 2016 Oct 4. PMID 27717842